CLINICAL TRIAL: NCT03467451
Title: Rétrospective Evaluation of the Performance and the Safety of the Endoscopic Mucosectomy With Anchorage of the Tip of the Loop
Brief Title: Rétrospective Evaluation of the Performance and the Safety of the Endoscopic Mucosectomy With Anchorage
Status: Completed | Type: Observational
Sponsor: Hôpital Edouard Herriot (Other)
Responsible Party: Principal Investigator, Jean Christophe Saurin, Professor, Société Française d'Endoscopie Digestive
Other Study IDs: Mucosectomy with anchorage
Record Dates: First submitted 2018-03-09; First posted 2018-03-16 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Polyps of Colon
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic Mucosectomy — Endoscopic Mucosectomy with anchorage of the tip of the loop

SUMMARY:
This safe and simple technique without extra cost would allow us to improve R0 resection ratio and so decrease relapses and the time between two different exams

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Other rectal or colic résections from 10 to 30 mm into the past

Exclusion Criteria:

* Colitis, Crohn Disease or Ulcerative Colitis
* Intense fibrosis under the lesion

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Both male and female over 18 years old with other rectal or colic résections from 10 to 30 mm into the past
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Measure the proportion of R0 resections of anchored mucosectomies from 10 to 30 mm colon and rectum lesions | One year

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu Pioche, Principal Investigator — Hôpital Edouard Herriot